CLINICAL TRIAL: NCT02176512
Title: Relative Oral Bioavailability of 80 mg Telmisartan / 12.5 mg HCTZ Fixed Dose Combination Compared With Its Monocomponents in Healthy Subjects. A 4 Period Cross-over, Open, Randomized, Replicate Design Study.
Brief Title: Telmisartan/Hydrochlorothiazide (HCTZ) Fixed Dose Combination Compared to Its Monocomponents in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 502.136
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Hydrochlorothiazide

ARMS (2):
- Sequence 1 (Experimental): four treatment periods:
  1. Treatment A
  2. Treatment B
  3. Treatment B
  4. Treatment A
  Interventions: Drug: BIBR 277 SE and HCTZ; Drug: BIBR 277 SE; Drug: HCTZ
- Sequence 2 (Active Comparator): four treatment periods:
  1. Treatment B
  2. Treatment A
  3. Treatment A
  4. Treatment B
  Interventions: Drug: BIBR 277 SE and HCTZ; Drug: BIBR 277 SE; Drug: HCTZ

INTERVENTIONS:
Drug: BIBR 277 SE and HCTZ — Treatment A - fixed dose combination
Drug: BIBR 277 SE — Treatment B - Monocomponent
Drug: HCTZ — Treatment B -Monocomponent

SUMMARY:
Study to demonstrate the bioequivalence of telmisartan and HCTZ administered as fixed dose combination in comparison to the single unit formulations

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by results of screening
* Signed written informed consent in accordance with GCP (Good Clinical Practice) and local legislation
* Age ≥ 18 and ≤ 45 years
* Broca ≥ - 20% and ≤ + 20%

Exclusion Criteria:

* Any findings of the medical examination (including blood pressure, pulse rate and ECG and laboratory value) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastro-intestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Supine blood pressure at screening of systolic ≤ 110 mmHg and diastolic ≤ 60 mmHg
* History of orthostatic hypotension, fainting spells or blackouts
* Hypersensitivity to Telmisartan and/or HCTZ and/or related classes of drugs
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Use of any drugs which might influence the results of the trial (≤ 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (≤ 2 months prior to administration or during the trial)
* Smoker (≥ 10 cigarettes or ≥ 3 cigars or ≥ 3 pipes/day)
* Inability to refrain from smoking on study days
* Known alcohol abuse
* Known drug abuse
* Blood donation (≤ 1 month prior to administration)
* Excessive physical activities (≤ 5 days prior to administration)
* For female subjects:

  * Pregnancy
  * Positive pregnancy test
  * No adequate contraception
  * Inability to maintain this adequate contraception during the whole study period
  * Lactation period

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 1998-09; Primary Completion 1998-10 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (total area under the plasma drug concentration-time curve from time zero to infinity) | up to 96 hours post-dose
Cmax (maximum drug plasma concentration) | up to 96 hours post-dose
Amount of Hydrochlorothiazide (HCTZ) excreted in urine over 48 hours (Ae(0-48h)) | 0-6, 6-12, 12-24, 24-32, 32-48 hours post-dose

SECONDARY OUTCOMES:
tmax (time to achieve Cmax) | up to 96 hours post-dose
t1/2 (apparent terminal elimination half-life) | up to 96 hours post-dose
CLtot/f (total clearance of a drug from plasma, divided by bioavailability) | up to 96 hours post-dose
MRTtot (mean time of residence of drug molecules in the body) | up to 96 hours post-dose
Vz/f (apparent volume of distribution during terminal phase) | up to 96 hours post-dose
Number of patients with adverse events | Up to 62 days